CLINICAL TRIAL: NCT05239598
Title: A Phase II, Randomized Trial to Test the Effect of Povidone-iodine 0.5% as Mouthwash/Gargle on SARS-CoV-2 Load (COVID 19) as an Adjuvant Infection Control Measure in Dental Practice
Brief Title: Povidone-Iodine Oral Rinse Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Avrio Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 849386
Record Dates: First submitted 2022-02-14; First posted 2022-02-15 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Mouthwashes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Povidone-iodine 0.5% antiseptic mouth rinse (Experimental): Subjects will be asked to rinse/gargle one time with 10 mL of Povidone-iodine 0.5% antiseptic mouth rinse for 30 seconds.
  Interventions: Drug: Mouth rinse
- Placebo (Placebo Comparator): Subjects will be asked to rinse/gargle one time with 10 mL of placebo mouth rinse for 30 seconds.
  Interventions: Drug: Mouth rinse

INTERVENTIONS:
Drug: Mouth rinse — Subjects will be asked to rinse/gargle one time with 10 mL of assigned mouth rinse for 30 seconds.

SUMMARY:
This study is a two-arm, randomized, 2-phase study. Phase I will be double blinded clinical trial of the safety and efficacy of an antiseptic mouthwash solution on reducing SARS-CoV-2 load in COVID 19+ adult individuals. Phase II is designed as an open label trial, and all subjects will receive the active mouthwash.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide informed consent prior to initiation of study procedures.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged 18 years and older.
4. Clinical diagnosis of COVID-19 infection confirmed with a positive point of care test.
5. Confirmed diagnosis within 5 days of baseline visit (within 5 days of COVID-19 test) and at least one clinical COVID-19 symptom [*Signs and symptoms of COVID-19 present at illness onset vary, but over the course of the disease, most people will experience the following: fever or chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste of smell, sore throat, congestion or runny nose, nausea or vomiting and diarrhea.]
6. Presents with a minimum of six natural teeth.
7. Ability to rinse/gargle with study products.
8. Not using mouth rinse/gargling solutions at the time of enrollment.
9. Not taking antimicrobial medications (antibacterial, antiviral, antibiotics, including hydroxychloroquine) at time of enrollment.
10. Ability to participate in the study and come to site during Phase I of the study for collection of swabs and saliva.
11. Willing to use an acceptable method of birth control throughout duration of the study. Acceptable methods include hormonal contraceptives, barrier methods, abstinence, or other effective methods approved by the PI.
12. If continuing to Phase II of the trial, ability to continue using study products for 1 week (+ 3 days). (Participants do not have to agree to participate in Phase II in order to participate in Phase I.)
13. If continuing to Phase II of the trial, agree to receive text messages/phone calls containing questionnaires regarding compliance and use of study product, and reminders, able to complete virtual follow-up study visit for collection of outcomes data.

Exclusion Criteria:

1. Individuals receiving antiviral medications
2. Pregnant or breastfeeding women (for premenopausal women of childbearing potential, pregnancy status to be confirmed through a urine pregnancy test during the study visit)
3. Inability to comply with study protocol
4. Having an allergy to any of the study mouthwash ingredients
5. Having any thyroid condition.
6. Presents with a current suspicious oral lesion at the examiner's discretion, and/or currently undergoing radiation therapy for head or neck cancer, and/or has received radiation therapy to the head or neck (including radioactive iodine therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Corby, DDS, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from 2/7/2022 to 7/7/2022. Primary recruitment was through the University of Pennsylvania testing sites, community testing sites, and community partners. We also placed flyers/advertisements within our hospitals and dental clinics, including our community health centers outside the school, and relevant social media pages.
Groups:
- Povidone-iodine 0.5% Antiseptic Mouth Rinse: Subjects were asked to rinse/gargle one time with 10 mL of Povidone-iodine 0.5% antiseptic mouth rinse for 30 seconds.
  Mouth rinse: Subjects were asked to rinse/gargle one time with 10 mL of assigned mouth rinse for 30 seconds.
- Placebo: Subjects were asked to rinse/gargle one time with 10 mL of placebo mouth rinse for 30 seconds.
  Mouth rinse: Subjects were asked to rinse/gargle one time with 10 mL of assigned mouth rinse for 30 seconds.
Period: Phase I
Arm/Group | Povidone-iodine 0.5% Antiseptic Mouth Rinse | Placebo
Started | 21 | 19
Completed | 21 | 19
Not Completed | 0 | 0
Period: Phase II (Open Label)
Arm/Group | Povidone-iodine 0.5% Antiseptic Mouth Rinse | Placebo
Started | 37 | 0
Completed | 35 | 0
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Povidone-iodine 0.5% Antiseptic Mouth Rinse | Placebo | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.6 (11.4) | 32.4 (12.3) | 31.5 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 5 | 7 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 20 | 19 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 7 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 10 | 15
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 2 | 0 | 2
(PCR Saliva) Ct Viral target Means (SD) at baseline [Mean (Standard Deviation); unit: Cycle Threshold] — Higher mean "Cycle Threshold" represent lower SARS-Co-V-2 load, this is represented by CT RT-PCR values on an inverse correlation.
  PCR TRESHOLD: COVID-Seq requires specimen with Cycle Threshold values <30 to proceed - Cycle Threshold value >30 is considered negative. [Quick SARS-CoV-2 rRT-PCR Kit (Zymo Research, Cat. No. R3011)]. Three participants had non-evaluable baseline Cycle Threshold-values and were not included in analysis. Population: 3 subjects (2 randomized to Povidone-iodine arm, and 1 randomized to Placebo) had non-evaluable baseline Cycle Threshold values and were not included in analysis.
  Cycle Threshold
    number analyzed (Participants) | 19 | 18 | 37
    (all) | 26.6 (4.7) | 25.1 (5.6) | 25.9 (5.1)
[Oropharyngeal Swab] Log10 Antigens [Median (Inter-Quartile Range); unit: Log10 Copies/mL] — Antigen analysis detects the viral antigen, or protein components of the virus (it can be associated with "Acute infection").
  Microbubbling Digital Assay: TARGET N proteins from SARS-CoV-2 viruses. Output is the signal level that is given by nucleocapsid antigen in the samples when bound to antibodies.
  Log10 Copies/mL | 4.3 [3.9 to 5.2] | 4.2 [3.7 to 5.2] | 4.3 [3.8 to 5.2]
[Nasal Swab] Log10 Antigens [Median (Inter-Quartile Range); unit: Log10 Copies/mL] — In the context of the study, the nasal antigen data was used to validate infectivity, as the site was not treated. Data show all subjects had strong antigen signals from nasal swab samples at all timepoints.
  Antigen analysis detects the viral antigen, or protein components of the virus (it can be associated with "Acute infection").
  Microbubbling Digital Assay: TARGET N proteins from SARS-CoV-2 viruses. Output is the signal level that is given by nucleocapsid antigen in the samples when bound to antibodies.
  Log10 Copies/mL | 6.2 [5.4 to 6.5] | 6.3 [6.0 to 6.5] | 6.2 [5.6 to 6.5]

OUTCOME MEASURES:

1. Primary Outcome: [PCR Saliva] Percent Change From Baseline Ct Viral Targets
Description: The primary endpoint is the percentage reduction of SARS-Co-V-2 load in saliva at 60 minutes (post-intervention) compared to baseline between the PVP-I mouthwash versus the placebo mouthwash. For this outcome, Cycle Threshold is a proxy for SARS-Co-V-2 load. A positive percent change from baseline Cycle Threshold indicates a decrease from baseline SAR-Co-V2.
  [Quick SARS-CoV-2 rRT-PCR Kit (Zymo Research, Cat. No. R3011)].
Time Frame: 60 minutes after intervention
Population: Participants were randomized to Povidone-iodine or Placebo (saline) in a 1:1 ratio. Three participants had non-evaluable baseline Cycle Threshold-values and one value was missing at 60 minutes so they were excluded from the analysis of the outcome.
Measure: Mean (95% Confidence Interval); unit: % Change from Baseline Cycle Threshold
Groups:
- Povidone-iodine 0.5% Antiseptic Mouth Rinse: Subjects were asked to rinse/gargle one time with 10 mL of Povidone-iodine 0.5% antiseptic mouth rinse for 30 seconds. Saliva samples were obtained at baseline and at 5, 30, 60 minutes post intervention.
- Placebo: Subjects were asked to rinse/gargle one time with 10 mL of placebo (saline) mouth rinse for 30 seconds. Saliva samples were obtained at baseline and at 5, 30, 60 minutes post intervention.
Arm/Group | Povidone-iodine 0.5% Antiseptic Mouth Rinse | Placebo
Number analyzed (Participants) | 19 | 17
% Change from Baseline Cycle Threshold | 5.8 [0.8 to 10.7] | 1.3 [-6.2 to 8.8]
Statistical Analysis 1: Comparison: Povidone-iodine 0.5% Antiseptic Mouth Rinse vs Placebo; Test type: Superiority; p = 0.287, t-test, 2 sided; Mean Difference (Net) = 4.5, 95% CI 2-sided [-4.0 to 13.0]

2. Secondary Outcome: [PCR Saliva] Percent Change From Baseline Cycle Threshold at 5 and 30 Minutes Post Intervention
Description: The secondary endpoints are the percentage reduction of SARS-Co-V-2 load in saliva at 5 and 30 minutes (post-intervention) compared to baseline between the PVP-I mouthwash versus the placebo mouthwash. For this outcome, Cycle Threshold is a proxy for SARS-Co-V-2 load. A positive percent change from baseline Cycle Threshold indicated a decrease from baseline SARS-Co-V-2.
Time Frame: 5 and 30 minutes post-intervention
Population: Participants were randomized to Povidone-iodine or Placebo (saline) in a 1:1 ratio. Three participants had non-evaluable baseline Ct-values so were excluded from the analysis of these secondary outcomes.
Measure: Mean (95% Confidence Interval); unit: % Change from Baseline Cycle Threshold
Arm/Group | Povidone-iodine 0.5% Antiseptic Mouth Rinse | Placebo
Number analyzed (Participants) | 19 | 18
% Change from Baseline Cycle Threshold
  5 minutes post intervention | 3.3 [-2.1 to 8.7] | 1.7 [-3.0 to 6.3]
  30 minutes post intervention | 2.0 [-2.5 to 6.5] | -0.6 [-7.6 to 6.5]
Statistical Analysis 1: Comparison: Povidone-iodine 0.5% Antiseptic Mouth Rinse vs Placebo; 5 minutes post intervention; Test type: Superiority; p = 0.625, t-test, 2 sided; Mean Difference (Net) = 1.7, 95% CI 2-sided [-5.2 to 8.6]
Statistical Analysis 2: Comparison: Povidone-iodine 0.5% Antiseptic Mouth Rinse vs Placebo; 30 minutes post intervention; Test type: Superiority; p = 0.526, t-test, 2 sided; Mean Difference (Net) = 2.5, 95% CI 2-sided [-5.5 to 10.5]

3. Other Pre Specified Outcome: [Oropharyngeal Swab] Percent Change From Baseline Log10 Antigens
Description: The secondary endpoints are the percentage reduction in SARS-Co-V-2 antigens obtained from oropharyngeal swab at 5, 30 and 60-minutes (post-intervention) compared to baseline within each treatment group.
Time Frame: 5, 30, and 60 minutes post intervention
Population: Participants were randomized to Povidone-iodine or Placebo (saline) in a 1:1 ratio.
Measure: Median (Inter-Quartile Range); unit: % Change from Baseline Median Log10
Groups:
- Povidone-iodine 0.5% Antiseptic Mouth Rinse: Subjects were asked to rinse/gargle one time with 10 mL of Povidone-iodine 0.5% antiseptic mouth rinse for 30 seconds. Oropharyngeal swab samples were obtained at baseline and at 5, 30, 60 minutes post intervention.
- Placebo: Subjects were asked to rinse/gargle one time with 10 mL of placebo (saline) mouth rinse for 30 seconds. Oropharyngeal swab samples were obtained at baseline and at 5, 30, 60 minutes post intervention.
Arm/Group | Povidone-iodine 0.5% Antiseptic Mouth Rinse | Placebo
Number analyzed (Participants) | 21 | 19
% Change from Baseline Median Log10
  5 minutes post intervention | 0.04 [-4.2 to 8.1] | -2.4 [-6.5 to -0.9]
  30 minutes post intervention | 5.4 [-10.7 to 18.6] | -6.6 [-10.1 to -2.2]
  60 minutes post intervention | -4.9 [-15.2 to 17.5] | -8.6 [-22.3 to -3.9]
Statistical Analysis 1: Comparison: Povidone-iodine 0.5% Antiseptic Mouth Rinse; Povidone-iodine: 5 minutes Post-Intervention; Test type: Superiority; p = 0.511, Signed Rank; Median Difference (Net) = 0.04, 95% CI 2-sided [-4.2 to 8.1]
Statistical Analysis 2: Comparison: Povidone-iodine 0.5% Antiseptic Mouth Rinse; Povidone-iodine: 30 minutes post-intervention; Test type: Superiority; p = 0.408, Signed Rank; Median Difference (Net) = 5.4, 95% CI 2-sided [-10.7 to 18.6]
Statistical Analysis 3: Comparison: Povidone-iodine 0.5% Antiseptic Mouth Rinse; Povidone-iodine: 60 minutes post-intervention; Test type: Superiority; p = 0.907, Signed Rank; Median Difference (Net) = -4.9, 95% CI 2-sided [-15.2 to 17.5]
Statistical Analysis 4: Comparison: Placebo; Placebo: 5 minutes post intervention; Test type: Superiority; p = 0.008, Signed Rank; Median Difference (Net) = -2.4, 95% CI 2-sided [-6.5 to -0.9]
Statistical Analysis 5: Comparison: Placebo; Placebo: 30 minutes post-intervention; Test type: Superiority; p = 0.080, Signed Rank; Median Difference (Net) = -6.6, 95% CI 2-sided [-10.1 to -2.2]
Statistical Analysis 6: Comparison: Placebo; Placebo: 60 minutes post-intervention; Test type: Superiority; p = 0.001, Signed Rank; Median Difference (Net) = -8.6, 95% CI 2-sided [-22.3 to -3.9]

4. Other Pre Specified Outcome: [Nasal Swab] Log10 Antigens
Description: In the context of the study, the antigen data was used to validate infectivity, as this site was not treated. The pre-specified outcomes are the percentage reduction in SARS-Co-V-2 antigens obtained from nasal swab at 5, 30 and 60-minutes (post-intervention) compared to baseline within each treatment group.
Time Frame: 5, 30, 60 minutes post intervention
Population: Participants were randomized to Povidone-iodine or Placebo (saline) in a 1:1 ratio.
Measure: Median (Inter-Quartile Range); unit: % Change from Baseline Log10 Antigens
Groups:
- Povidone-iodine 0.5% Antiseptic Mouth Rinse: Subjects were asked to rinse/gargle one time with 10 mL of Povidone-iodine 0.5% antiseptic mouth rinse for 30 seconds. Nasal swab samples were obtained at baseline and at 5, 30, 60 minutes post intervention.
- Placebo: Subjects were asked to rinse/gargle one time with 10 mL of placebo (saline) mouth rinse for 30 seconds. Nasal swab samples were obtained at baseline and at 5, 30, 60 minutes post intervention.
Arm/Group | Povidone-iodine 0.5% Antiseptic Mouth Rinse | Placebo
Number analyzed (Participants) | 21 | 19
% Change from Baseline Log10 Antigens
  5 minutes post intervention | 3.1 [-2.2 to 5.8] | -4.1 [-7.1 to 0.7]
  30 minutes post intervention | 1.8 [-2.3 to 6.9] | -0.7 [-9.4 to 2.0]
  60 minutes post intervention | 1.5 [-3.1 to 6.8] | -3.6 [-7.7 to 4.0]
Statistical Analysis 1: Comparison: Povidone-iodine 0.5% Antiseptic Mouth Rinse; Povidone-iodine 5 minutes post-intervention; Test type: Superiority; p = 0.212, Signed Rank; Median Difference (Net) = 3.1, 95% CI 2-sided [-2.2 to 5.8]
Statistical Analysis 2: Comparison: Povidone-iodine 0.5% Antiseptic Mouth Rinse; Povidone-iodine 30 minutes post-intervention; Test type: Superiority; p = 0.334, Signed Rank; Median Difference (Net) = 1.8, 95% CI 2-sided [-2.3 to 6.9]
Statistical Analysis 3: Comparison: Povidone-iodine 0.5% Antiseptic Mouth Rinse; Povidone-iodine 60 minutes post-intervention; Test type: Superiority; p = 0.269, Signed Rank; Median Difference (Net) = 1.5, 95% CI 2-sided [-3.1 to 6.8]
Statistical Analysis 4: Comparison: Placebo; Placebo 5 minutes post-intervention; Test type: Superiority; p = 0.026, Signed Rank; Median Difference (Net) = -4.1, 95% CI 2-sided [-7.1 to -0.7]
Statistical Analysis 5: Comparison: Placebo; Placebo 30 minutes post-intervention; Test type: Superiority; p = 0.182, Signed Rank; Median Difference (Net) = -0.7, 95% CI 2-sided [-9.4 to 2.0]
Statistical Analysis 6: Comparison: Placebo; Placebo 60 minutes post-intervention; Test type: Superiority; p = 0.353, Signed Rank; Median Difference (Net) = -3.6, 95% CI 2-sided [-7.7 to 4.0]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time of informed consent was obtained until 7 (for non-serious AEs) or 30 days (for SAEs) after the last day of study participation. Note, no SAEs were reported.
Groups:
- Phase II - Open Label: All subjects in Phase II will be asked to use the Povidone-iodine 0.5% mouth rinse for 1 week. They will be asked to rinse/gargle with 10mL mouthwash for 30 seconds 4 times per day for 1 week.
Arm/Group | Povidone-iodine 0.5% Antiseptic Mouth Rinse | Placebo | Phase II - Open Label
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/37
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 4/37
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Povidone-iodine 0.5% Antiseptic Mouth Rinse (N=40) | Placebo (N=40) | Phase II - Open Label (N=37)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Tingling Tongue (General disorders) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Our findings suggest that RT-PCR quantification of Ct viral targets present some limitations but can be of clinical utility. RT-PCR methods are inherently quantitative, and reproducible during repeated clinical sampling over a short time period. A limitation of our study was that changes in viral targets (RT-PCR) was determined after a one-time use of the mouthwash; prolonged use might yield better efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT05239598/Prot_SAP_001.pdf